CLINICAL TRIAL: NCT00233298
Title: A Study of the Function of Hormones Present In Taste Buds
Status: Completed | Type: Observational
Sponsor: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999905254; 05-AG-N254
Record Dates: First submitted 2005-10-03; First posted 2005-10-05 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2015-01-02

CONDITIONS: Diabetes; Obesity; Pre-Diabetes; Metabolic Syndrome
Keywords: Hypoglycemia; Blood Sugar; Blood Glucose Level; Insulin Sensitivity; Metabolism; Type 2 Diabetes; Healthy
MeSH Terms: conditions — Diabetes Mellitus; Obesity; Glucose Intolerance; Metabolic Syndrome; Hypoglycemia; Insulin Resistance; Diabetes Mellitus, Type 2

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The purpose of this study is to find out whether the hormones in the taste buds are affected by tasting and eating food, and also whether these hormone levels are affected by an increase in body weight or type 2 diabetes.

DETAILED DESCRIPTION:
Cephalic phase of insulin secretion is regulated by autonomic and endocrine responses to food-related sensory stimulation such as sight, smell, and taste. Human taste perception comprises of at least five distinct qualities: bitterness, saltiness, sourness, sweetness, and umami, the sensation elicited by glutamate, commonly found in protein (meat, fish, and legumes) and flavor enhancer such as monosodium glutamate (MSG).

Both the sweet and umami taste stimuli had been shown to illicit cephalic-phase insulin release in rats. Oral sensory stimulation in human with modified sham feeding (MSF where food is smelled, chewed, but not swallowed) had been shown to enhance insulin release during the cephalic phase, lower postprandial glucose level, and improve glucose tolerance in healthy subjects. The loss of pre-absorptive insulin response has been shown to impair glucose tolerance. Furthermore, patients with type 2 diabetes and their first degree relatives had been shown to have impairment of sweet taste.

Recently, glucagon-like peptide-1 (GLP-1) and peptide YY (PYY) have been found in the taste cells located in the taste buds of mice (unpublished data). These new findings raise several interesting questions of whether strict tasting of food without ingestion may stimulate secretion of GLP-1 and PYY from the taste cells, whether their secretion is involved in the afferent input of the cranial nerves, and whether this secretion is impaired in obesity and in patients with pre-diabetes or type 2 diabetes. We also want to investigate whether different tastants, such as sweet versus umami, and different food contents such as percent fat versus carbohydrate compositions, would elicit different hormonal responses.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Males or females age 20 to 50
  2. body weight > 50 kg (110 pounds)
  3. Group A

     1. BMI < 25 kg/m(2)
     2. healthy
  4. Group B

     1. BMI greater than or equal to 30 kg/ m(2)
     2. healthy
  5. Group C

     1. Pre-diabetes
     2. Pre-diabetes is defined as having either impaired fasting glucose (IFG) (fasting plasma glucose (FPG) greater than or equal to100 mg/dl but < 126 mg/dl) and/or impaired glucose tolerance (IGT) (2-hour OGTT glucose greater than or equal to140 mg/dl but < 200 mg/dl).
     3. BMI greater than or equal to 30 kg/m(2)
  6. Group D

     1. Type 2 diabetes (on diet or oral agents management only except for thiazolidinediones)
     2. Type 2 diabetes is defined as FPG 126 mg/dl and/or 2-hour OGTT glucose

        200
     3. BMI greater than or equal to 30 kg/m(2)
  7. Screening laboratory evaluations with no significant abnormal results:

     1. comprehensive metabolic panel
     2. complete blood count with differential and platelets
     3. fasting plasma glucose < 100 mg/dl for healthy groups only (Group A and B)
     4. 2-hour 75-gram OGTT glucose < 140 mg/dl for healthy groups only (Group A and B)
     5. Negative pregnancy test for women of child-bearing potential
  8. Able to complete an informed consent

EXCLUSION CRITERIA:

1. Pregnancy (pregnancy has been shown to be associated with decrease in insulin sensitivity
2. Group A and B subjects cannot have FPG greater than or equal to 100 mg/dl or 2-hr OGTT greater than or equal to 140 mg/dl
3. Group D subjects cannot have FPG > 240 mg/dl during the screening visit
4. Group D subjects cannot have their morning fasting finger-stick glucose > 240 mg/dl during the 5 days (3 days for glucophage) prior to the visit when their oral hypoglycemic agent(s) are discontinued
5. Subjects with type 2 diabetes on insulin therapy
6. Hematocrit < 36% for women and < 38% for men
7. Peanut allergy
8. Presence of other medical conditions that could affect glucose homeostasis
9. Use of medications known to impair glucose homeostasis (i.e., amiloride shown to inhibit certain taste responses in hamsters)
10. History of liver or renal disease
11. History of gastrointestinal or endocrine disorders except for treated hypo- or hyperthyroidism
12. Long-term glucocorticoid use (over one month), or other immunosuppressive agents within the past 5 years

Ages: 12 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 225 (Actual)
Dates: Start 2005-05-26; Study Completion 2015-01-02

PRIMARY OUTCOMES:
Whether CLP-1 and PYY are involved in the cephalic phase response during feeding | 12 months
Differences in response among healthy, healthy obese, pre-diabetic or 3 diabetes | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Josephine M Egan, M.D., Principal Investigator — National Institute on Aging (NIA)
Locations (1):
- National Institute of Aging, Clinical Research Unit, Baltimore, Maryland, United States

REFERENCES:
- [Background] Ahren B. Autonomic regulation of islet hormone secretion--implications for health and disease. Diabetologia. 2000 Apr;43(4):393-410. doi: 10.1007/s001250051322. PMID 10819232
- [Background] Lindemann B. Taste reception. Physiol Rev. 1996 Jul;76(3):719-66. doi: 10.1152/physrev.1996.76.3.719. PMID 8757787
- [Background] Niijima A, Togiyama T, Adachi A. Cephalic-phase insulin release induced by taste stimulus of monosodium glutamate (umami taste). Physiol Behav. 1990 Dec;48(6):905-8. doi: 10.1016/0031-9384(90)90247-2. PMID 2087524